CLINICAL TRIAL: NCT02146586
Title: Cooperative International Neuromuscular Research Group (CINRG) Clinical Evaluator Outcomes Reliability Study
Brief Title: Clinical Evaluator Outcomes Reliability Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Cooperative International Neuromuscular Research Group (Network)
Responsible Party: Sponsor
Other Study IDs: CNMC0713
Record Dates: First submitted 2014-05-14; First posted 2014-05-26 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-02

CONDITIONS: Dystrophinopathies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Dystrophinopathies
- Gold Standard Clinical Evaluators (GS-CEs)
- Sites Clinical Evaluators (CEs)

SUMMARY:
This study outlines structured Clinical Evaluator (CE) testing techniques that are proposed to be implemented across all sites participating in the Cooperative International Neuromuscular Research Group (CINRG) research studies. The study will determine if the selected techniques are reliable and reproducible across the CINRG network by evaluating the reliability and reproducibility of the measures between CEs

ELIGIBILITY:
Dystrophinopathy Participant Inclusion Criteria:

* Site confirmed genetic diagnosis of a dystrophinopathy
* Aged 6 years and older
* Able to transfer to testing table
* Able to walk 10 meters without an assistive device

Dystrophinopathy Participant Exclusion Criteria:

* Investigator assessment of inability to comply with protocol assessments
* Participants who have attention deficient disorder or other cognitive conditions that may limit attention span to perform protocol assessments

Min Age: 6 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Dystrophinopathies (Duchenne Muscular Dystrophy and Becker Muscular Dystrophy)
Sampling Method: Non-Probability Sample
Enrollment: 55 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Clinical Evaluator Assessments | One time visit
  The following assessments are conducted by certified physical therapists: Anthropometrics, goniometry, Brooke upper extremity and Vignos lower extremity scales, Performance Upper Limb Scale (PULS), North Star Ambulatory Assessment (NSAA), Six Minute Walk Test (6MWT), time to rise from floor, time to stand from a chair, time to climb four stairs, time to walk/run 10 meters, 9 Hole Peg Test (9HPT), Quantitative Muscle Tests (QMT), Manual Muscle testing (MMT), Force Vital Capacity (FVC), Force Expiratory Volume (FEV1), Maximum Inspiratory Pressure (MIP), Maximum Expiratory Pressure (MEP), Peak Expiratory Flow Rate (PEFR) and Peak Cough Flow (PCF).
  The reliability of these commonly used measurements is fundamental to clinical research, our ability to have confidence in the data we collect and our ability to draw rational conclusions from the data.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Morgenroth, MS, CGC, Principal Investigator — Children's National Research Institute; Tina Duong, MPT, Principal Investigator — Stanford University